CLINICAL TRIAL: NCT01126775
Title: Neuro-Prävention im Rahmen Des Interventionsprojektes INVADE-2 Systematische Prävention Bei Hochrisikopatienten für Schlaganfall Und vaskulär (Mit)Bedingte Demenz: Identifizierung Und Behandlung Von Stummen Hirninfarkten.
Brief Title: Neuro-Prävention im Rahmen Des Interventionsprojektes INVADE-2 (Follow-up Studie)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: INVADE gGmbH (Other)
Responsible Party: Sponsor
Other Study IDs: INV-1006-Gna-1000-I
Record Dates: First submitted 2010-05-18; First posted 2010-05-20 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2013-01

CONDITIONS: Stroke; Dementia
Keywords: Systematic prevention, stroke, vascular dementia, silent strokes, cerebral microangiopathy.
MeSH Terms: conditions — Stroke; Dementia; Dementia, Vascular; Cerebral Small Vessel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- group non-high-risk
- group high risk

SUMMARY:
"Silent" strokes are more frequent than clinical apparent strokes and can be detected noninvasively by MRI-investigations of the brain. Persons with silent strokes have a considerably increased risk for clinical apparent strokes as well as for the development of dementia. Intention of the study is the detection of silent strokes and microbleedings by standardized cranial MRI in 1000 participants (500 high-risk and 500 low-risk persons for cerebrovascular accidents) after a standardized neurological and neuropsychological examination. Results will be the base of early detection and early preventive strategies of cerebrovascular accidents in high-risk persons.

In the course of a systematic follow-up examination without MRI the same 1000 patients (500 high-risk and 500 low-risk persons for cerebrovascular accidents) will be reinvited to the sites. In addition to the standardized neurological and neuropsychological examinations a surrogate parameter of nephropathy, microalbumin, will be examined as this parameter could be helpful in forecasting cerebral microangiopathy. The clinical investigation will be expanded by several tests in order to assess symptoms of cerebral microangiopathy.

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent for NPV-2
* ongoing participation in INVADE-2
* completed participation in Neuroprävention study (NPV-1)

Exclusion Criteria:

* not completed Neuroprävention study (Drop-out)
* disagreement of notification of incidental findings
* lack of capacity to consent of study participant
* lack of willingness to cooperate of study participant

Min Age: 55 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 1000 participants of INVADE-2-study ("Intervention project on cerebrovascular diseases and dementia in the district of Ebersberg, Bavaria")
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2012-04; Primary Completion 2013-11 (Estimated)

PRIMARY OUTCOMES:
In the group of high-risk persons the percentage of silent strokes detected by MRI of the brain is significantly higher than in the group of non-high-risk persons. | 4/2012 until 11/2013

SECONDARY OUTCOMES:
Detection of silent strokes by MRI in more than 10% of all subjects and diagnostic and therapeutic procedures refinancable near-term and in relation to long-term-consequences | 4/2012 until 11/2013
Detection of microbleedings by MRI in more than 10% of all subjects | 4/2010 until 11/2011

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - Praxis Dr. Briesenick u. Dr. Förstner, Baldham, Bavaria
  - Praxis Dr. Gnahn u. Dr. Klein, Ebersberg, Bavaria

REFERENCES:
- [Background] Scherpinski U, Bickel H, Gnahn H, Forstl H, Conrad B, Sander D. [Intervention project on cerebrovascular diseases and dementia in the Ebersberg district (INVADE): rationale and design]. Nervenarzt. 2002 Dec;73(12):1199-204. doi: 10.1007/s00115-002-1443-8. German. PMID 12486573